CLINICAL TRIAL: NCT05080153
Title: The Effects of Vitamin Supplementation Containing L-Methylfolate (Ocufolin® Forte) on Retinal Venous Pressure and Homocysteine Plasma Levels in Patients With Glaucoma
Brief Title: Effect of Vitamin Supplementation in Glaucoma Patients
Status: Completed | Type: Observational
Sponsor: Devogelaere Vision (Other)
Responsible Party: Principal Investigator, Thibaut Devogelaere, Dr T Devogelaere, MD, FEBO, Devogelaere Vision
Other Study IDs: 151119-OcF
Record Dates: First submitted 2021-10-05; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Glaucoma; Homocysteinemia; Elevated Retinal Venous Pressure; Abnormal Steady State Pattern Electroretinography
Keywords: glaucoma; homocysteine plasma levels; L-methylfolate; ophthalmodynamometry; retinal venous pressure (RVP); steady state pattern electroretinography
MeSH Terms: conditions — Glaucoma; Homocysteinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Ocufolin forte — start of ocufolin forte 1 dd after RVP measurement, till 90 tablets are finished (3 months)

SUMMARY:
The impact of targeted vitamin supplementation on retinal venous pressure (RVP) and steady state pattern ERG (SSpERG) in patients with RVP 15mmHg or more above intra-ocular pressure (IOP) and serum homocystein 12µmol/l or more, with signs of progression in spite of adequate IOP control, as evidenced by SSpERG abnormality with or without structural progression or visual field progression,

DETAILED DESCRIPTION:
Provided the inclusion criteria were met, RVP measurement was repeated, and a 1 capsule/day regimen of Ocufolin® forte was subsequently carried out for a duration of 3 months, after which repeat measurements of IOP, SSpERG, and RVP were performed, along with dilated fundoscopy. .

ELIGIBILITY:
Inclusion Criteria:

* glaucoma and/or ocular vascular disease in at least on eye
* abnormal SSpERG
* RVP measured using an ophthalmodynamometer at least 15 mmHg higher than intra-ocular pressure (IOP),
* fasting serum Hcy level > 12 µmol/l
* stable and well-controlled IOP (with or without IOP-lowering treatment)

Exclusion Criteria:

* starting other systemic or ocular medications with potential impacts on RVP within a month before entering the study or during the course of the study
* starting or changing the dosage of other medications with potential impact on SSpERG within 3 months before entering the study or during the course of the study
* non-adherence to the follow-up schedule
* inability to perform a proper RVP measurement using ophthalmodynamometry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with glaucoma and/or ocular vascular disease with signs of progression in spite of well controlled IOP and elevated RVP, with fasting serum Hcy level > 12 µmol/l
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
RVP effect | 3 months
  measurement of RVP lowering effect
SSpERG effect | 3 months
  measurement of improvement of SSpERG

CONTACTS AND LOCATIONS:
Overall Officials: Thibaut Devogelaere, MD, FEBO, Principal Investigator — Vision Devogelaere
Locations (1):
- Devogelaere Vision, Oudenburg, Belgium

IPD SHARING:
Plan to Share IPD: No